CLINICAL TRIAL: NCT05327907
Title: Establishment of Scoring Model for Early Diagnosis and Differential Diagnosis of Intrahepatic Cholangiocarcinoma
Brief Title: Establishment of Scoring Model for Early and Differential Diagnosis of Intrahepatic Cholangiocarcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Jinan Central Hospital (Other); Shandong Provincial Hospital (Other Government); Jinan Military General Hospital (Other)
Responsible Party: Principal Investigator, Yanjing Gao, Clinical Professor, Qilu Hospital of Shandong University
Other Study IDs: 202135719-Qilu
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Intrahepatic Cholangiocarcinoma
Keywords: Intrahepatic cholangiocarcinoma; Hepatocellular carcinoma; radiomics; nomogram
MeSH Terms: conditions — Cholangiocarcinoma; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Training cohort: Training cohort consists of the patients diagnosed with intrahepatic cholangiocarcinoma who collected from January 2010 to July 2021 retrospectively.
- Internal validation cohort: Internal validation cohort consists of the intrahepatic cholangiocarcinoma patients who enrolled from September 2021 of Qilu Hospital prospectively.
- External validation cohort: External validation cohort consists of the intrahepatic cholangiocarcinoma patients who enrolled from September 2021 of Shandong Province Hospital, Jinan Military General Hospital and Jinan Central Hospital prospectively.

SUMMARY:
The purpose of this study is to develop and validate a radiological nomogram including radiological characteristics, clinical risk factors, and medical history. And we aim to establish a noninvasive method for the diagnosis of intrahepatic cholangiocarcinoma (ICC), and to construct a differential diagnosis model for ICC and hepatocellular carcinoma (HCC) with higher sensitivity and accuracy.

DETAILED DESCRIPTION:
In recent years, the incidence and mortality of intrahepatic cholangiocarcinoma (ICC) have been increasing worldwide. Due to the different treatment options for hepatocellular carcinoma (HCC) and ICC, accurate differential diagnosis is critical for subsequent treatment of patients. However, because of their similar CT image enhancement patterns, they are easily misdiagnosed by clinicians, leading to an incorrect treatment. Based on the above research background, our objective is to establish a noninvasive method for the diagnosis of ICC and and to construct a differential diagnosis model for ICC and HCC with higher sensitivity and accuracy.

ELIGIBILITY:
Inclusion Criteria:

1. patients with pathological confirmation of ICC or HCC,
2. CT was performed less than 15 days before surgery,
3. Patients with complete clinical data.

Exclusion Criteria:

1. history of other tumors,
2. Metastatic liver cancer,
3. Patients received preoperative chemotherapy or radiotherapy,
4. Image quality analysis is not ideal.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical data of patients in hospitals in the past 10 years were retrospectively collected. Pathological database from September 2010 to July 2021 was searched. Patients with definite pathological diagnosis of ICC or HCC were determined as the training group, and patients from September 2021 to September 2023 were prospectively collected as the validation group.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-11-22 (Actual); Primary Completion 2023-02-22 (Estimated); Study Completion 2023-05-22 (Estimated)

PRIMARY OUTCOMES:
Accuracy | through study completion, up to 2 years
  The golden standard is the pathological biopsy.Compare the accuracy of the noninvasive model with the pathological biopsy.
sensitivity | through study completion, up to 2 years
  Sensitivity of noninvasive model for diagnosis of intrahepatic cholangiocarcinoma.
specificity | through study completion, up to 2 years
  Specificity of noninvasive model for diagnosis of intrahepatic cholangiocarcinoma.

CONTACTS AND LOCATIONS:
Overall Officials: Yanjing Gao, PhD.MD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology,Qilu Hospital,Shandong University, Jinan, Shandong, China